CLINICAL TRIAL: NCT03248297
Title: Azithromycin With or Without Amoxicillin to Prevent Peripartum Infection and Sepsis in Laboring High-risk Women: 3-Arm RCT
Brief Title: Antibiotic Prophlaxis for High-risk Laboring Women in Low Income Countries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alan Tita, Professor and Director, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHI UAB MISP # 54628
Record Dates: First submitted 2017-07-25; First posted 2017-08-14 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-03

CONDITIONS: Postpartum Sepsis; Postpartum Endometritis; Postpartum Fever
MeSH Terms: conditions — Puerperal Infection | interventions — Azithromycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azithromycin and amoxicillin placebo (Experimental): Patients in this arm will receive 1 gram oral azithromycin as a single dose and amoxicillin placebo.
  Interventions: Drug: Azithromycin; Drug: Placebo
- Azithromycin + amoxicillin (Experimental): Patients in this arm will receive 1 gram oral azithromycin and 2 grams oral amoxicillin in a single dose.
  Interventions: Drug: Azithromycin and amoxicillin
- Usual Care (Placebo Comparator): This arm will consist of routine care at the clinical sites (which is usually no antibiotic). They will receive placebo (for azithromycin) and placebo (for amoxicillin)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin tablet
  Arms: Azithromycin and amoxicillin placebo
Drug: Azithromycin and amoxicillin — azithromycin and amoxicillin
  Other Names: azithromycin, amoxicillin
  Arms: Azithromycin + amoxicillin
Drug: Placebo — Placebo tablet
  Arms: Azithromycin and amoxicillin placebo; Usual Care

SUMMARY:
This study, performed over a course of 3 years in 5 collaborating hospitals in Cameroon, Africa, will randomize 750 women in labor with prolonged rupture of membranes ≥ 8 hours or prolonged labor ≥ 18 hours to identical oral regimens of 1 gram of azithromycin, 1 gram of azithromycin+2 grams of amoxicillin or placebo. Women will be followed to ascertain maternal infectious outcomes and perinatal outcomes.

DETAILED DESCRIPTION:
This 3-arm study is a large randomized clinical trial designed to evaluate the comparative effectiveness and safety of single dose oral azithromycin or combined azithromycin+amoxicillin compared to placebo for the prevention of peripartum infections and sepsis in laboring women. We have previously shown the effectiveness of azithromycin for extended spectrum antibiotic prophylaxis in addition to the standard cephalosporin alone for reduction of post-cesarean infections. In LICs, the fraction of maternal infection and sepsis from cesarean delivery is minimal. Therefore, it is necessary to evaluate strategies aimed at reducing these morbidities in women who have vaginal births. There is an increased risk of infection in women who have prolonged labor or prolonged rupture of membranes. Drawing from our findings with azithromycin-based extended antibiotic prophylaxis for cesarean delivery, we propose to adapt the intervention and evaluate a single oral dose of azithromycin (with or without oral amoxicillin) to prevent maternal peripartum infection and sepsis. This study, performed over a course of 3 years in 5 collaborating hospitals in Cameroon, Africa, will randomize 750 women in labor with prolonged rupture of membranes ≥ 8 hours or prolonged labor ≥18 hours to 1 gram of oral azithromycin, 1 gram of azithromycin+2 grams of amoxicillin, compared to usual care (placebo). Women will be followed to ascertain maternal infectious outcomes and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 37 weeks' viable singleton or twin gestation in labor planning a vaginal delivery with

  1. Prolonged membrane rupture (≥8 hours) or
  2. Prolonged labor (≥18 hours).

Exclusion Criteria:

* Clinical chorioamnionitis or any other active bacterial infection (e.g. pyelonephritis, pneumonia, abscess) at time of randomization: because standard antibiotic therapy for these conditions may confound trial intervention.
* Allergy to azithromycin or amoxicillin
* Plan for cesarean delivery prior to enrollment
* Fetal demise or major congenital anomaly: Major congenital anomalies may confound assessment of neonatal outcomes and every attempt will be made up front to exclude them from randomization. However, some unrecognized fetal anomalies may inevitably be randomized. These will not be excluded post-randomization from the primary (maternal outcome) analysis; they will be taken into consideration in the secondary analyses of neonatal outcomes.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 756 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tita, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Cameroon Baptist Convention Health Services, Bamenda, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] ASHP Therapeutic Guidelines on Antimicrobial Prophylaxis in Surgery. American Society of Health-System Pharmacists. Am J Health Syst Pharm. 1999 Sep 15;56(18):1839-88. doi: 10.1093/ajhp/56.18.1839. No abstract available. PMID 10511234
- [Background] Tita ATN, Boggess K, Saade G. Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. N Engl J Med. 2017 Jan 12;376(2):182. doi: 10.1056/NEJMc1614626. No abstract available. PMID 28076707
- [Background] WHO Recommendations for Prevention and Treatment of Maternal Peripartum Infections. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK327079/ PMID 26598777
- [Derived] Subramaniam A, Ye Y, Mbah R, Mbunwe DM, Pekwarake S, Bunwi EY, Fondzeyuf A, Ngong MG, Dionne-Odom J, Harper LM, Jauk VC, Carlo WA, Halle-Ekane G, Szychowski JM, Tih P, Tita AT. Single Dose of Oral Azithromycin With or Without Amoxicillin to Prevent Peripartum Infection in Laboring, High-Risk Women in Cameroon: A Randomized Controlled Trial. Obstet Gynecol. 2021 Nov 1;138(5):703-713. doi: 10.1097/AOG.0000000000004565. PMID 34619734

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Started | 253 | 253 | 250
Completed | 253 | 253 | 250
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care | Total
Number analyzed (Participants) | 253 | 253 | 250 | 756
Age, Customized [Mean (Standard Deviation); unit: years] | 27.2 (5.3) | 26.4 (5.6) | 26.0 (5.3) | 26.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 253 | 250 | 756
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 253 | 253 | 250 | 756
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 253 | 253 | 250 | 756
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Gestational age at Randomization [Mean (Standard Deviation); unit: Weeks] | 39.4 (1.5) | 39.2 (1.4) | 39.2 (1.4) | 39.3 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Composite Peripartum Infection or Death
Description: Maternal peripartum infection including chorioamnionitis, endometritis, wound infection/abscess, sepsis, and death
Time Frame: Up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 15 | 17 | 24

2. Secondary Outcome: Number of Participants Who Experienced Pyelonephritis
Description: Other Infections
Time Frame: Up to hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 2 | 2 | 3

3. Secondary Outcome: Number of Participants Who Experienced Breast Infection
Description: Other infections
Time Frame: Up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 2 | 0 | 0

4. Secondary Outcome: Number of Participants Who Experienced Other Infection
Description: Includes Hepatitis B, thyroid infection, vaginal infection, viral infection, leg cellulitis, unknown abdominal infection,malaria
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 4 | 3 | 1

5. Secondary Outcome: Number of Participants Who Experienced Fever
Description: Any fever higher than 38C
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 22 | 21 | 28

6. Secondary Outcome: Number of Participants Who Experienced Hypothermia
Description: Any hypothermia less than 36C
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 9 | 11 | 15

7. Secondary Outcome: Number of Participants Who Needed PP Antibiotic
Description: Any postpartum antibiotic
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 18 | 18 | 26

8. Secondary Outcome: Number of Participants Who Experienced Transfusion
Description: Blood transfusion
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 8 | 3 | 4

9. Secondary Outcome: Number of Participants Who Experienced Stillbirth
Description: Any stillbirth
Time Frame: delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 1 | 0 | 1

10. Secondary Outcome: Length of Stay
Description: Length of stay in days
Time Frame: up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
days | 3.7 (2.0) | 3.7 (2.2) | 3.8 (3.1)

11. Secondary Outcome: Number of Participants Who Experienced a Clinic Visit
Description: Clinic visit after discharge
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 13 | 7 | 10

12. Secondary Outcome: Number of Participants Who Experienced a Maternal Readmission
Description: Maternal readmission
Time Frame: up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
Number analyzed (Participants) | 253 | 253 | 250
Participants | 11 | 4 | 5

ADVERSE EVENTS:
Time Frame: up to 6 weeks after delivery
Arm/Group | Azithromycin and Amoxicillin Placebo | Azithromycin + Amoxicillin | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/253 | 0/250
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/253 | 0/250
Other Adverse Events (participants affected / at risk) | 0/253 | 0/253 | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT03248297/Prot_SAP_000.pdf